CLINICAL TRIAL: NCT06025071
Title: Efficacy and Safety of Residual Inflammatory Risk-Guided Low-dose Colchicine Therapy in Elderly Patients With Multivessel Coronary Artery Disease: A Multicenter Randomized Controlled Trial
Brief Title: Residual Inflammatory Risk-Guided colcHicine in Elderly Trial
Acronym: RIGHT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xueyan Zhao, Chief physician, M.D., FACC, FESC, Doctoral supervisor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-GSP-GG-40
Record Dates: First submitted 2023-06-02; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Percutaneous Coronary Intervention; Multivessel Coronary Artery Disease; Elderly Patients; C-Reactive Protein
Keywords: multivessel coronary artery disease; percutaneous coronary intervention; elderly patients; colchicine; high sensitive-C reactive protein; efficacy and safety
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Open-label, Two-arm, Randomized, Superiority Trial
Who Masked: Outcomes Assessor
Masking Description: This is an open-lable study. But while the study is in progress, the grouping information is masked from outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine group (Experimental): Drug: Colchicine; Dosage form: Tablets; Dosage: 0.5mg; Frequency: Once daily; Duration: From randomization to one-year follow-up is completed.
  Interventions: Drug: colchicine
- Control group (No Intervention): No intervention

INTERVENTIONS:
Drug: colchicine — Dosage form: Tablets; Dosage: 0.5mg; Frequency: Once daily; Duration: From randomization to one-year follow-up is completed.
  Arms: Colchicine group

SUMMARY:
The goal of this clinical trial is to compare low-dose colchicine (0.5 mg Once Daily) with no specific intervention in selected elderly patients (60-80 years old) with residual inflammatory risk (hs-CRP≥ 2mg/L) and multivessel coronary artery disease. The main questions it aims to answer are:

* Whether the intervention is effective in reducing ischemic events
* Whether the intervention is effective in reducing inflammatory biomarkers' level
* Whether the intervention is safe for elderly patients

Participants will be randomized to receive low-dose colchicine (0.5 mg Once Daily) or no specific intervention for one year. Patients enrolled should complete one-year follow-up in the form of clinic visit or telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-80 years old
* Baseline plasma hs-CRP≥2 mg/L
* Hospitalized patients with coronary artery disease with multi-vessel lesions (multi-vessel lesions are defined as at least 2 major epicardial coronary arteries with ≥50% stenosis in their main branch diameter confirmed by coronary CT or coronary angiography, with or without left main artery disease)
* Patients with myocardial ischemia-related symptoms or objective evidence are successfully treated with PCI, and the condition is relatively stable
* Received standard drug therapies based on their condition at baseline (including antiplatelet, lipid-lowering, blood pressure control, blood glucose control, and other treatments recommended by guidelines)
* Subjects or legal representatives have signed informed consent.

Exclusion Criteria:

* Patients who have acute myocardial infarction within 30 days
* Patients who have taken colchicine and have a clear history of allergy or intolerance
* Patients with renal insufficiency, eGFR <30 ml/min/1.73 m^2 (calculated by MDRD formula) or blood creatinine levels exceeding 2 times the upper normal limit
* Patients with cirrhosis, chronic active hepatitis, liver function impairment (alanine aminotransferase exceeding 3 times the upper normal limit or total bilirubin exceeding 2 times the upper normal limit) or cholestasis
* Patients with a known history of hypomyelodysplasia
* Patients with heart failure (NYHA Class III-IV) or severe valvular disease
* Patients with concomitant neoplastic or cancer disease
* Patients with chronic obstructive pulmonary disease or other chronic pulmonary disease
* Patients with poorly controlled disease, such as current cardiogenic shock, hemodynamic instability, heart failure (NYHA Class III-IV), left ventricular ejection fraction less than 35%, recent stroke (within the past 3 months), or any other condition in which the investigator believes that participation in this study puts the patient at risk
* Patients with inflammatory bowel disease (Crohn's disease or ulcerative colitis) or chronic diarrhea
* Patients with hemoglobin less than 115 g/L, white blood cell count less than 4.0*10^9/L, or platelet count less than 110*10^9/L
* Patients are currently using or plan to begin chronic systemic steroid therapy (oral or intravenous) during the study period (topical or inhaled steroids are allowed)
* Patients with acute inflammation or viral infection
* Female patients who are currently pregnant, planning to become pregnant, or breastfeeding

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | From randomization to occurence of first event, assessed up to one year
  Composite events including cardiovascular death, spontaneous (nonprocedural) myocardial infarction, ischemia-driven coronary revascularization, and ischemic stroke

SECONDARY OUTCOMES:
Cardiovascular death | From randomization to occurence of first event, assessed up to one year
  Number of participants with cardiovascular death.
Spontaneous (nonprocedural) myocardial infarction | From randomization to occurence of first event, assessed up to one year
  Number of participants with spontaneous (nonprocedural) myocardial infarction.
Ischemia-driven coronary revascularization | From randomization to occurence of first event, assessed up to one year
  Number of participants with ischemia-driven coronary revascularization.
Ischemic stroke | From randomization to occurence of first event, assessed up to one year
  Number of participants having had a ischemic stroke.
Change of hs-CRP | From randomization to treatment at one month and one year
  Change of hs-CRP comparing to the baseline
Change of white blood cell count | From randomization to treatment at one month and one year
  Change of white blood cell count comparing to the baseline
Change of neutrophil count | From randomization to treatment at one month and one year
  Change of neutrophil count comparing to the baseline
Change of monocyte count | From randomization to the end of treatment at one year
  Change of monocyte count comparing to the baseline

OTHER OUTCOMES:
Nausea | From randomization to treatment at one month and one year
  Treatment-related adverse events as nausea
Vomiting | From randomization to treatment at one month and one year
  Treatment-related adverse events as vomiting
Diarrhea | From randomization to treatment at one month and one year
  Treatment-related adverse events as diarrhea
Abdominal pain | From randomization to treatment at one month and one year
  Treatment-related adverse events as abdominal pain
Muscle pain | From randomization to treatment at one month and one year
  Treatment-related adverse events as muscle pain
Neuritis | From randomization to treatment at one month and one year
  Treatment-related adverse events as neuritis
Rash | From randomization to treatment at one month and one year
  Treatment-related adverse events as rash
Gout | From randomization to treatment at one month and one year
  Treatment-related adverse events as gout
Hospitalization for infections | From randomization to treatment at one month and one year
  Treatment-related adverse events as hospitalization for infections
New tumors | From randomization to treatment at one month and one year
  Treatment-related adverse events as new tumors
Blood pressure | From randomization to treatment at one month and one year
  Both systolic and diastolic blood pressure
Heart rate | From randomization to treatment at one month and one year
White blood cell count | From randomization to treatment at one month and one year
Neutrophil count | From randomization to treatment at one month and one year
Monocyte count | From randomization to treatment at one month and one year
Hematocrit | From randomization to treatment at one month and one year
Hemoglobin level | From randomization to treatment at one month and one year
Platelet count | From randomization to treatment at one month and one year
Alanine aminotransferase | From randomization to treatment at one month and one year
Aspartate aminotransferase | From randomization to treatment at one month and one year
Gamma-glutamyltransferase | From randomization to treatment at one month and one year
Total bilirubin | From randomization to treatment at one month and one year
Direct bilirubin | From randomization to treatment at one month and one year
Serum albumin | From randomization to treatment at one month and one year
Total serum protein | From randomization to treatment at one month and one year
Serum creatinine | From randomization to treatment at one month and one year
Blood urea nitrogen | From randomization to treatment at one month and one year
Creatine Kinase | From randomization to treatment at one month and one year

CONTACTS AND LOCATIONS:
Overall Officials: Xueyan Zhao, M.D., Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Diseases, CAMS & PUMC
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, CAMS & PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No